CLINICAL TRIAL: NCT01402271
Title: Phase IB-II, Open Label, Multicenter Feasibility Study of Pazopanib in Combination With Paclitaxel and Carboplatin in Patients With Platinum-Refractory/Resistant Ovarian, Fallopian Tube or Peritoneal Carcinoma
Brief Title: Pazopanib Hydrochloride, Paclitaxel, and Carboplatin in Treating Patients With Refractory or Resistant Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-55092; EU-21119; 2010-024077-39 (EudraCT Number)
Record Dates: First submitted 2011-07-23; First posted 2011-07-26 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; recurrent fallopian tube cancer; recurrent primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Paclitaxel

ARMS (2):
- pazopanib in combination with paclitaxel and carboplatin (Experimental): Phase I: Dose-escalation study of pazopanib in combination with paclitaxel and carboplatin given weekly in a group of patients with platinum-refractory or -resistant ovarian, fallopian tube or peritoneal carcinoma Phase II: Paclitaxel 30 mg/m² and Carboplatin 2.0 AUC weekly for 18 courses PLUS Pazopanib 400 mg daily
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: pazopanib hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study
- Paclitaxel and carboplatin only (Active Comparator): Carboplatin AUC 2.7 and paclitaxel 60mg/m² weekly for 18 courses.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: pazopanib hydrochloride

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: pazopanib hydrochloride
Other: laboratory biomarker analysis
  Arms: pazopanib in combination with paclitaxel and carboplatin
Other: pharmacological study
  Arms: pazopanib in combination with paclitaxel and carboplatin

SUMMARY:
RATIONALE: Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of pazopanib hydrochloride when given together with paclitaxel and carboplatin in treating patients with refractory or resistant ovarian epithelial cancer, fallopian tube cancer, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose of pazopanib hydrochloride in combination with paclitaxel and carboplatin in patients with platinum-refractory or -resistant ovarian epithelial, fallopian tube, or peritoneal carcinoma. (Phase I)
* To determine the progression-free survival (PFS) at 1 year according to the RECIST 1.1 in these patients. (Phase II)

Secondary

* To determine the safety and adverse event profiles in these patients. (Phase I and phase II)
* To determine the pharmacokinetics (PK) of this regimen using intensive sampling. (Phase I)
* To determine if there is PK interaction (and if so, what kind of PK interaction) between carboplatin and paclitaxel as well as pazopanib hydrochloride. (Phase I)
* To determine the response rate (RR) in these patients. (Phase I)
* To determine and evaluate predictive biomarkers. (Phase I and phase II)
* To determine the RR, overall survival (OS), and PFS of these patients. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of carboplatin, paclitaxel, and pazopanib hydrochloride followed by a phase II randomized study.

* Phase I: Patients receive paclitaxel IV over 1 hour followed by carboplatin IV over 30 minutes on day 1. Patients also receive oral pazopanib hydrochloride* once daily on days 2-7. Treatment repeats every week for up to 18 courses**. Patients then continue to receive oral pazopanib hydrochloride once daily in the absence of disease progression or unacceptable toxicity.

NOTE: *Pazopanib hydrochloride is started in course 2 in order to evaluate the pharmacokinetic of paclitaxel and carboplatin prior to pazopanib hydrochloride administration.

* Phase II: Patients are stratified according to center, disease status (platinum-refractory vs -resistant) and number of prior lines of treatment (1 vs more than 1). Patients are randomized in a 2:1 ratio (arm II [experimental arm]: arm I [standard arm]) to 1 of 2 treatment arms.

  * Arm I (standard arm): Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Treatment repeats every week for up to 18 courses.
  * Arm II (experimental arm): Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Patients also receive oral pazopanib hydrochloride once daily on days 2-7. Treatment repeats every week for up to 18 courses**. Patients then continue to receive oral pazopanib hydrochloride once daily in the absence of disease progression or unacceptable toxicity.

NOTE: **After course 9, chemotherapy will be interrupted for 1 week.

Blood samples are collected from some patients periodically for pharmacokinetic and biomarker studies.

After completion of study treatment, patients are followed up at 3 weeks, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or peritoneal carcinoma

  * Recurrent disease
* Received at least 1 prior platinum treatment and developed platinum-refractory disease (i.e., progression within 4 weeks of platinum administration) or platinum-resistant disease (i.e., progression within 6 months after the last platinum dose)

  * There is no restriction on the number of prior lines of treatment
  * Non-platinum treatment is allowed after proven platinum-resistance or -refractory disease
* Evaluable (measurable or nonmeasurable) disease according to RECIST version 1.1 criteria
* Patients with refractory disease on weekly paclitaxel and carboplatin regimen are excluded (phase II only)
* No known gastrointestinal intraluminal metastatic lesions with risk of bleeding
* No known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* No known brain metastases or leptomeningeal disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100 x 10^9/L
* PT, aPTT, or INR ≤ 1.2 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN*
* ALT and AST ≤ 2.5 times ULN*
* Serum creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance ≥ 50 mL/min
* Urine protein creatinine ratio < 1 OR 24-hour urine protein < 1 g
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study therapy
* No other prior primary or recurrent malignancies treated within the past 2 years except for completely resected non-melanomatous skin carcinoma or successfully treated carcinoma in situ of the skin or uterine cervix
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs similar or related to paclitaxel, carboplatin, and pazopanib hydrochloride
* Able to receive infusions of paclitaxel and carboplatin
* Able to swallow pazopanib hydrochloride tablets
* No unstable or serious condition (e.g., uncontrolled infection requiring systemic therapy)
* No history of any of the following cardiovascular conditions within the past 6 months:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic peripheral vascular disease
  * NYHA class III-IV congestive heart failure
* LVEF > 50% as assessed by ultrasound or MUGA scan, if clinically indicated
* No inadequately controlled hypertension (SBP ≥ 140 mm Hg or DBP ≥ 90 mm Hg)

  * Initiation or adjustment of blood pressure medication is permitted prior to the study entry
* No prolonged corrected QT interval (QTc) defined as > 480 msecs using Bazett formula
* No history of cerebrovascular accident within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Pulmonary embolism
  * Untreated deep venous thrombosis (DVT)

    * Patients with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* No evidence of active bleeding or bleeding diathesis
* No clinically significant gastrointestinal (GI) tract abnormalities that may increase the risk for GI bleeding including, but not limited to, any of the following:

  * Active peptic ulcer disease
  * Inflammatory bowel disease (e.g., ulcerative colitis or Crohn disease)
* No history of bowel obstruction (excluding postoperative (i.e. within 4 weeks post surgery)) during the whole prior history of the patient, or other GI condition with increased risk of perforation such as clear infiltration into the rectosigmoid, colon or small bowel.
* No clinically significant GI abnormalities that may affect absorption of investigational product including, but not limited to, any of the following:

  * Malabsorption syndrome
  * Major resection of stomach or small bowel
* No hemoptysis in excess of 2.5 mL (one-half teaspoon) within 8 weeks prior to first dose of study drug
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No trauma within the past 28 days
* No prior non-healing wounds, fracture, or ulcer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No ongoing toxicity from prior anticancer therapy > grade 1 and/or that is progressing in severity, except for alopecia and ≤ grade 2 peripheral neuropathy
* No cardiac angioplasty or stenting within the past 6 months
* No coronary artery bypass graft surgery within the past 6 months
* At least 14 days since prior radiotherapy, surgery, or tumor embolization , chemotherapy, immunotherapy, biologic therapy, investigational therapy, or hormonal therapy (28 days for drugs with a longer half-life)
* At least 14 days since prior (28 days for drugs with a longer half-life) and no concurrent prohibited medications
* At least 28 days since prior major surgery (procedures such as catheter placement and diagnostic endoscopic procedures are not considered to be major)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-07; Primary Completion 2019-05-15 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of pazopanib hydrochloride, carboplatin, and paclitaxel (phase I)
Progression-free survival according to RECIST 1.1 at 1 year (phase II)

SECONDARY OUTCOMES:
Pharmacokinetics of pazopanib, carboplatin, and paclitaxel (phase I)
Safety and tolerability according to CTCAE 4.0 (phase I and phase II)
Response rate (phase I and phase II)
Predictive biomarkers (phase I and phase II)
Overall survival (phase II)
Age-related subanalysis for toxicity and efficacy (cut-off 65 years old) (phase II)

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (5):
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - U.Z. Gasthuisberg, Leuven
  - C.H.U. Sart-Tilman, Liège
  - Centre Hospitalier Regional De La Citadelle, Liège
  - ZNA Jan Palfijn, Merksem
- Netherlands (2):
  - Radboud University Medical Center Nijmegen, Nijmegen
  - Erasmus MC, Rotterdam
- Spain (2):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona
  - Hospital Clínico Universitario San Carlos, Madrid